CLINICAL TRIAL: NCT02507193
Title: Fibular Fixation in Ankle Fractures: a Randomized-Controlled Trial Comparing Plating Versus Intramedullary Nailing
Brief Title: Fibular Fixation in Ankle Fractures:Plate Verses Nail.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Paula J. Harriott, Clinical Research Coordinator, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.037.04.
Record Dates: First submitted 2015-06-03; First posted 2015-07-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2018-10

CONDITIONS: Distal Fibula Fracture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open reduction internal fixation(ORIF) (Active Comparator): This surgical intervention is performed using a plate and screws.Under general anesthesia, an incision is made at the site of the break or injury, and the fracture is carefully re-aligned . The plate and screws are installed, and the incision is closed with staples or stitches. Synthes and Stryker plate and screws will be used.
  Interventions: Procedure: Open reduction internal fixation
- Intermedullary (IM) Nail (Active Comparator): This surgical intervention is performed using an intermedullary nail. Under general anesthesia, an incision is made at the site of the break or injury, and the fracture is carefully reduced. The nail in inserted through the medullary canal after proper imaging for accurate placement. The incision is closed with staples or stitches. Acumed fibula nail will be used.
  Interventions: Procedure: Intermedullary Nail

INTERVENTIONS:
Procedure: Open reduction internal fixation — An incision is made at the site of the break or injury, and the fracture is carefully re-aligned . The plate and screws are installed, and the incision is closed with staples or stitches. Synthes and Stryker plate and screws will be used.
  Other Names: ORIF
  Arms: Open reduction internal fixation(ORIF)
Procedure: Intermedullary Nail — An incision is made at the site of the break or injury, and the fracture is carefully reduced. The nail in inserted through the medullary canal after proper imaging for accurate placement. The incision is closed with staples or stitches. Acumed fibula nail will be used.
  Arms: Intermedullary (IM) Nail

SUMMARY:
The primary objective of this study will be to evaluate the functional outcome of patients who present with a distal fibula fracture who were treated with either intermedullary nail (IMN) fixation or plate fixation.

DETAILED DESCRIPTION:
The primary objective of this study will be to evaluate the functional outcome of patients who present with a distal fibula fracture who were treated with either intermedullary nail (IMN) fixation or plate fixation. This objective will be accomplished using the Olerud-Molander score, a commonly accepted functional outcome score used to evaluate patients post-operatively who have undergone foot and ankle procedures. It is a survey that evaluates patient reported outcomes including pain, stiffness, swelling, stair climbing, running, jumping, squatting, use of supports, and work/activities of daily living (ADL) level. It does not involve physician-measured outcomes. The best possible score is a total of 100. Patients will be given a form to complete throughout follow-up and be utilized for data analysis. Functional outcome will be analyzed with regards to type of fracture, gender, cause of fracture, and affected side to determine if these factors are responsible for any difference.

ELIGIBILITY:
Inclusion Criteria:

* Distal fibula fracture
* Pilon fractures
* Open fractures
* Ipsilateral foot

Exclusion Criteria:

* Weber A distal fibula fractures
* Pathologic fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Functional outcome using the Olerud-Molander score. | One year.
  The Olerud-Molander score is as assessment of symptoms after ankle fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. Koval, MD, Study Director — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States